CLINICAL TRIAL: NCT03448679
Title: Serum Albumin, Colloid Osmotic Pressure and Endothelial Damage in Patients With End Stage Liver Disease Undergoing Orthotopic Liver Transplantation. A Retrospective Data Analysis.
Brief Title: Albumin, COP and Endothelial Damage in Patients With ESLD Undergoing OLT
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, PD Peter Faybik, MD, Assoc.Prof. PD MD, Medical University of Vienna
Other Study IDs: 2026/2015
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Transplant-Related Disorder
Keywords: glycocalyx; serum albumin; orthotopic liver transplantation; colloid osmotic pressure; endothelial dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum-samples for detection of syndecan-1 concentration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study the correlation between colloid osmotic pressure, albumin and the loss of vascular integrity in terms of endothelial dysfunction in patients with ESLD undergoing OLT and its impact on the perioperative course, as well as on morbidity and mortality.

DETAILED DESCRIPTION:
Patients suffering from end-stage liver disease (ESLD) are critically ill. Still, therapeutic options are limited, no organ replacement procedure is available and orthotopic liver transplantation remains the unique therapy of choice.

ESLD is associated with a myriad of comorbidities, and is characterized by imbalances in the acid-base- status, coagulopathy, metabolic disorders and activation of the pro-inflammatory cascade. ESLD represents a state of generalized systemic inflammation subsequently leading to endothelial dysfunction and capillary leak syndrome, potentially culminating in end-organ dysfunction.

Furthermore, patients with ESLD suffer from reduced regenerative and synthetic capacity/ability, which is reflected by the serum albumin deficiency. Serum albumin is the most important plasma protein, is produced exclusively in the liver, and houses various physiological functions: it owns immunological, immuno-modulating and anti-inflammatory properties, transport capacities, as well as detoxifying qualities. However, the most well known property of human serum albumin is maintaining the colloid osmotic pressure (COP). In the healthy individual, serum albumin is responsible for 75% up to 80% of the COP, whereas in the critically ill, the percentage proportion drops down to 17%. The COP itself accounts for the regulation and distribution of the plasma volume and is therefore essential in maintaining the vascular stability and integrity. Additionally, the endothelial glycocalyx is necessary in the context of safeguarding the endothelial function and regulating the vascular permeability. The glycocalyx covers the endothelium luminally and its core component is the heparan sulfate proteoglycan, syndecan-1. Under various clinical conditions, like ischemia/reperfusion, inflammation, sepsis, shock, major surgery, hypervolemia, degradation to the glycocalyx may happen. These pathophysiological circumstances may lead to loss of the endothelial integrity and consecutively to capillary-leak syndrome causing a loss of albumin and fluid extravasation/shifts. Various clinical and experimental studies could show that global, as well as regional ischemia and the subsequent reperfusion-phase, both lead to glycocalyx-shedding, in terms of increased syndecan-1 plasma levels. Furthermore, a previous study from our study group clearly detected increased syndecan-1 plasma levels in patients with ESLD as surrogate parameter of glycocalyx degradation mirroring the state of chronic inflammation in this patient population.

Nevertheless, a clear correlation between colloid osmotic pressure, albumin and the loss of vascular integrity in state of endothelial dysfunction has not been studied before in patients with ESLD undergoing OLT.

ELIGIBILITY:
Inclusion Criteria:

* Child B/C Cirrhosis
* patients, who undergo the first OLT

Exclusion Criteria:

* re-transplant
* pregnancy
* inoperability

Ages: 18 Years to 80 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18 years and 80 years suffering from Child B/C Cirhhosis, who underwent OLT at the Medical University of Vienna in the period between 2014 and 2016.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-12-06 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

PRIMARY OUTCOMES:
syndecan-1 | 5 days
  marker for endothelial damage